CLINICAL TRIAL: NCT03838549
Title: Pre Pectoral Implant for Immediate Breast Reconstruction Using Single Port Endoscopy in Prophylactic Indication
Acronym: MRIMOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Association la Montpellier Reine a du Cœur (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL18_0244; UF 7672 (Other: UH Montpellier)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Genetic Predisposition; Breast Cancer
Keywords: Prophylactic Surgical Procedure; Subcutaneous Mastectomy; Endoscopy; Breast Reconstruction; Breast Implants
MeSH Terms: conditions — Genetic Predisposition to Disease; Breast Neoplasms | interventions — Prophylactic Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- implant for breast reconstruction (Experimental): 20 patients female with genetic risk for breast cancer and who ask for prophylactic mastectomy. They will have a prophylactic mastectomy with immediate breast reconstruction
  Interventions: Procedure: Prophylactic mastectomy with immediate breast reconstruction

INTERVENTIONS:
Procedure: Prophylactic mastectomy with immediate breast reconstruction — It is an endoscopic approach for prophylactic mastectomy using an axillary single port

SUMMARY:
Implant-based reconstruction is currently the most common choice for mastectomy reconstruction. Whatever the choice of mastectomy incision, a scar remains on or near the breast volume. Current techniques involve partial or total coverage of the implant with the pectoralis major muscle, to prevent exposure or infection. The muscle dissection technique applied has functional and cosmetic consequences. In this study, an endoscopic approach will be evaluated. This new surgical technique, using a single-port endoscopic way, will put the scar is in the axillary area, away from the breast. The hypothesis is that this delocalized scar potentially reduces the risk of exposure and allows placement of the implant in the subcutaneous space, with no manipulation of the pectoralis major muscle.

DETAILED DESCRIPTION:
It s a practicability study, evaluating endoscopic approach for prophylactic mastectomy, using an axillary single port. Classic open surgery conversion rate, operative time, infectious rate, esthetical outcomes, and functional outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication for prophylactic uni or bilateral mastectomy (Genetic risk factors for breast cancer)
* Ask an immediate breast reconstruction during the surgery
* World Heath Organization score <3
* Glandular volume : french bra cup size A, B ou C
* Glandular ptosis <=2 (Classification and Algorithm for Treatment of Breast Ptosis)
* Contraception for woman of childbearing age and no pregnancy
* Valid Social Security
* Wrote consent

Exclusion Criteria:

* History of breast cancer surgery
* Breast cancer not operated on the side concerned by the prophylactic mastectomy
* Patient having had irradiant treatment
* Breast hypertrophy
* Smoking > 10 cigarette/day
* Body Mass Index > 30
* Large breast volume requiring prostheses > 500ml
* Chronic pulmonary obstructive gold 4
* ASA (Physical Status score of American Society of Anesthesiologists) > 3
* Chronic shoulder pain on the side to operate, or both shoulders
* History of abarticular pathology of the shoulder on the operating side
* Patient involvment in another clinical research
* Protected patient or unable to give consent
* Pregnant or breastfeeding woman
* Vulnerable person (Article L1121-6 of the Public Health Code)

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
success rate of total mastectomy | one day
  The total mastectomy is done by a scar in the axillary area, away from the breast, using single port endoscopy, with Implant base reconstruction in pre pectoral position.
  Complete excision of the gland by means of an incision on the axillary line, Installation of a definitive smooth prosthesis, Absence of conversion to a conventional approach, No skin necrosis

SECONDARY OUTCOMES:
Operative time | one day
  Duration of the prophylactic mastectomy with immediate breast reconstruction
Open surgery conversion rate | one day
  Open surgery conversion rate
Number of participants with an infection | 1 and 3 months after the prophylactic mastectomy
  Number of participants with early postoperative infection two months after the prophylactic mastectomy
Blood loss | one day
  Blood loss (milliliters) during the prophylactic mastectomy with immediate breast reconstruction
Number of participants with a local haematoma | Between the day of the prophylactic mastectomy and a month later
  Number of participants with a local haematoma caused by the prophylactic mastectomy with immediate breast reconstruction
Disunity of the scar | 1, 3, 6 and 12 months after the prophylactic mastectomy
  Number of patients with disunity of the scar after the prophylactic mastectomy
Exposure of the prosthesis | 1, 3, 6 and 12 months after the prophylactic mastectomy
  Number of patients with the prothesis exposed after the prophylactic mastectomy
Post-operative seromas after the prophylactic mastectomy | 1, 3, 6 and 12 months after the prophylactic mastectomy
  Number of patients with seromas after the prophylactic mastectomy
Complication rate of subcutaneous insufflation | 3 and 12 months after the prophylactic mastectomy
  Refractory induced hypercapnia: EtCO2 (expired fraction of CO2)> 45mmHg and refractory to ventilation ; second degree secondary burn
Skin case necrosis | 1, 3, 6 and 12 months after the prophylactic mastectomy
  The presence of skin case necrosis will be noted during all the visits after the surgery. It's severe if > 25%
Necrosis of areolo-nipple plaque | 1, 3, 6 and 12 months after the prophylactic mastectomy
  The presence of necrosis of areolo-nipple plaque will be noted during all the visits after the surgery.
Analogue visual scale (EVA) | 1, 3, 6 and 12 months after the prophylactic mastectomy
  The level of pain of the operated breasts will be self-assessed by the patient with EVA at 1, 3, 6, 12 months after the surgery. EVA is mesured between 0 and 10 (0: no pain ; 10: extremely intense pain)
Hospital stay | Through discharge from hospitalization, an average of 7 days
  The duration of hospitalization will be noted upon discharge from hospitalization
Aesthetic result | 3 and 12 months after the prophylactic mastectomy
  BREAST-Q© questionnaire Version 2.0 measure the quality of life and satisfaction among patients undergoing breast surgery. This questionnaire includes 6 modules: 1) Augmentation module, 2) Reduction/Mastectomy module, 3) Breast cancer: a) Mastectomy module, b) Reconstruction module, c) Breast reconstruction expectations module, d) Breast conserving therapy module.
  The conceptual framework of the modules is comprised of following two overarching themes (or domains): 1) Health-related quality of life and 2) Patient satisfaction. 1) Under each of these domains, there are six subthemes; Quality of life: 1) Psychosocial, 2) Physical and 3) Sexual well-being; and Patient satisfaction: 4) Satisfaction with Breasts, 5) Satisfaction with Outcome and 6) Satisfaction with care.
  Cf. https://qportfolio.org/wp-content/uploads/2020/BREAST-Q-USERS-GUIDE-V2.pdf for the response options.
Need for cosmetic reoperation | 3 and 12 months after the prophylactic mastectomy
  the need to use one or more lipomodelages
Shoulder function | 3 months after the prophylactic mastectomy
  Evaluation of the Constant score by a physiotherapist from the gynecology Department. The Constant score includes 5 items: Pain [0;5], Daily activity level [0;10], Level of work with the hand [0;10], Mobility [0;40] and Muscular force [0;25].
  The Constant score is mesured between 0 and 100. The higher the score, the fewer problems there are for the patient, 100 is the ideal score.
Life quality | 3 and 12 months after the prophylactic mastectomy
  Quality of life with an european quality of life scale (EQ-5D-3L). The EQ-5D-3L descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. Rated level can be coded as a number 1, 2, or 3, which indicates having no problems for 1, having some problems for 2, and having extreme problems for 3. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 33333 (having extreme problems in all dimensions).

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, Hérault, France

REFERENCES:
- [Background] Jakub JW, Peled AW, Gray RJ, Greenup RA, Kiluk JV, Sacchini V, McLaughlin SA, Tchou JC, Vierkant RA, Degnim AC, Willey S. Oncologic Safety of Prophylactic Nipple-Sparing Mastectomy in a Population With BRCA Mutations: A Multi-institutional Study. JAMA Surg. 2018 Feb 1;153(2):123-129. doi: 10.1001/jamasurg.2017.3422. PMID 28903167
- [Background] Colwell AS, Christensen JM. Nipple-Sparing Mastectomy and Direct-to-Implant Breast Reconstruction. Plast Reconstr Surg. 2017 Nov;140(5S Advances in Breast Reconstruction):44S-50S. doi: 10.1097/PRS.0000000000003949. PMID 29064921
- [Background] Muller T, Baratte A, Bruant-Rodier C, Bodin F, Mathelin C. Oncological safety of nipple-sparing prophylactic mastectomy: A review of the literature on 3716 cases. Ann Chir Plast Esthet. 2018 Jun;63(3):e6-e13. doi: 10.1016/j.anplas.2017.09.005. Epub 2017 Oct 10. PMID 29030030
- [Background] Casella D, Di Taranto G, Marcasciano M, Sordi S, Kothari A, Kovacs T, Lo Torto F, Cigna E, Ribuffo D, Calabrese C. Nipple-sparing bilateral prophylactic mastectomy and immediate reconstruction with TiLoop(R) Bra mesh in BRCA1/2 mutation carriers: A prospective study of long-term and patient reported outcomes using the BREAST-Q. Breast. 2018 Jun;39:8-13. doi: 10.1016/j.breast.2018.02.001. Epub 2018 Feb 18. PMID 29455110
- [Background] Miyake R, Kinoshita S, Shimada N, Uchida K, Takeyama H, Morikawa T. Preservation of the nipple-areola complex in skin-sparing mastectomy for early breast cancer. Surg Today. 2018 Jun;48(6):591-597. doi: 10.1007/s00595-018-1633-z. Epub 2018 Feb 21. PMID 29468434
- [Background] Co M, Chiu R, Chiu TM, Chong YC, Lau S, Lee YH, To HM, Kwong A. Nipple-Sparing Mastectomy and Its Application on BRCA Gene Mutation Carrier. Clin Breast Cancer. 2017 Dec;17(8):581-584. doi: 10.1016/j.clbc.2017.02.001. Epub 2017 Feb 14. PMID 28428099
- [Background] Ter Louw RP, Nahabedian MY. Prepectoral Breast Reconstruction. Plast Reconstr Surg. 2017 Nov;140(5S Advances in Breast Reconstruction):51S-59S. doi: 10.1097/PRS.0000000000003942. PMID 29064922
- [Background] Mitchell MP, Wagner J, Butterworth J. Subcutaneous implant-based breast reconstruction, a modern challenge in postmastectomy radiation planning. Pract Radiat Oncol. 2018 May-Jun;8(3):153-156. doi: 10.1016/j.prro.2017.09.001. Epub 2017 Sep 8. PMID 29233522
- [Background] Sbitany H, Piper M, Lentz R. Prepectoral Breast Reconstruction: A Safe Alternative to Submuscular Prosthetic Reconstruction following Nipple-Sparing Mastectomy. Plast Reconstr Surg. 2017 Sep;140(3):432-443. doi: 10.1097/PRS.0000000000003627. PMID 28574950
- [Background] Highton L, Johnson R, Kirwan C, Murphy J. Prepectoral Implant-Based Breast Reconstruction. Plast Reconstr Surg Glob Open. 2017 Sep 19;5(9):e1488. doi: 10.1097/GOX.0000000000001488. eCollection 2017 Sep. PMID 29062655
- [Background] Heidemann LN, Gunnarsson GL, Salzberg CA, Sorensen JA, Thomsen JB. Complications following Nipple-Sparing Mastectomy and Immediate Acellular Dermal Matrix Implant-based Breast Reconstruction-A Systematic Review and Meta-analysis. Plast Reconstr Surg Glob Open. 2018 Jan 12;6(1):e1625. doi: 10.1097/GOX.0000000000001625. eCollection 2018 Jan. PMID 29464161
- [Background] Glasberg SB. The Economics of Prepectoral Breast Reconstruction. Plast Reconstr Surg. 2017 Dec;140(6S Prepectoral Breast Reconstruction):49S-52S. doi: 10.1097/PRS.0000000000004051. PMID 29166348
- [Background] Kompatscher P. Endoscopic capsulotomy of capsular contracture after breast augmentation: a very challenging therapeutic approach. Plast Reconstr Surg. 1992 Dec;90(6):1125-6. doi: 10.1097/00006534-199212000-00049. No abstract available. PMID 1448521
- [Background] Lai HW, Chen ST, Chen DR, Chen SL, Chang TW, Kuo SJ, Kuo YL, Hung CS. Current Trends in and Indications for Endoscopy-Assisted Breast Surgery for Breast Cancer: Results from a Six-Year Study Conducted by the Taiwan Endoscopic Breast Surgery Cooperative Group. PLoS One. 2016 Mar 7;11(3):e0150310. doi: 10.1371/journal.pone.0150310. eCollection 2016. PMID 26950469
- [Background] Lai HW, Lin HY, Chen SL, Chen ST, Chen DR, Kuo SJ. Endoscopy-assisted surgery for the management of benign breast tumors: technique, learning curve, and patient-reported outcome from preliminary 323 procedures. World J Surg Oncol. 2017 Jan 11;15(1):19. doi: 10.1186/s12957-016-1080-5. PMID 28077134
- [Background] Lai HW, Lin SL, Chen ST, Kuok KM, Chen SL, Lin YL, Chen DR, Kuo SJ. Single-Axillary-Incision Endoscopic-Assisted Hybrid Technique for Nipple-Sparing Mastectomy: Technique, Preliminary Results, and Patient-Reported Cosmetic Outcome from Preliminary 50 Procedures. Ann Surg Oncol. 2018 May;25(5):1340-1349. doi: 10.1245/s10434-018-6383-z. Epub 2018 Feb 26. PMID 29484564
- [Background] Lai HW, Wu HS, Chuang KL, Chen DR, Chang TW, Kuo SJ, Chen ST, Kuo YL. Endoscopy-Assisted Total Mastectomy Followed by Immediate Pedicled Transverse Rectus Abdominis Musculocutaneous (TRAM) Flap Reconstruction: Preliminary Results of 48 Patients. Surg Innov. 2015 Aug;22(4):382-9. doi: 10.1177/1553350614546003. Epub 2014 Aug 12. PMID 25118202
- [Background] Leff DR, Vashisht R, Yongue G, Keshtgar M, Yang GZ, Darzi A. Endoscopic breast surgery: where are we now and what might the future hold for video-assisted breast surgery? Breast Cancer Res Treat. 2011 Feb;125(3):607-25. doi: 10.1007/s10549-010-1258-4. Epub 2010 Dec 3. PMID 21128113
- [Background] Wang Y, Wu JX, Guan S. A Technique of Endoscopic Nipple-Sparing Mastectomy for Breast Cancer. JSLS. 2017 Apr-Jun;21(2):e2017.00028. doi: 10.4293/JSLS.2017.00028. PMID 28684896
- [Background] Ng TB, Lee HM, Cheng CH, Wong CC. Study on the purification of growth hormone-like substance from pituitaries of the snake Ptyas mucosa. Prep Biochem. 1993 Aug;23(3):351-61. doi: 10.1080/10826069308544561. PMID 8361955
- [Background] Tukenmez M, Ozden BC, Agcaoglu O, Kecer M, Ozmen V, Muslumanoglu M, Igci A. Videoendoscopic single-port nipple-sparing mastectomy and immediate reconstruction. J Laparoendosc Adv Surg Tech A. 2014 Feb;24(2):77-82. doi: 10.1089/lap.2013.0172. Epub 2014 Jan 8. PMID 24401140
- [Background] Toesca A, Peradze N, Galimberti V, Manconi A, Intra M, Gentilini O, Sances D, Negri D, Veronesi G, Rietjens M, Zurrida S, Luini A, Veronesi U, Veronesi P. Robotic Nipple-sparing Mastectomy and Immediate Breast Reconstruction With Implant: First Report of Surgical Technique. Ann Surg. 2017 Aug;266(2):e28-e30. doi: 10.1097/SLA.0000000000001397. No abstract available. PMID 28692558
- [Background] Toesca A, Peradze N, Manconi A, Galimberti V, Intra M, Colleoni M, Bonanni B, Curigliano G, Rietjens M, Viale G, Sacchini V, Veronesi P. Robotic nipple-sparing mastectomy for the treatment of breast cancer: Feasibility and safety study. Breast. 2017 Feb;31:51-56. doi: 10.1016/j.breast.2016.10.009. Epub 2016 Nov 2. PMID 27810700
- [Background] Sarfati B, Struk S, Leymarie N, Honart JF, Alkhashnam H, Tran de Fremicourt K, Conversano A, Rimareix F, Simon M, Michiels S, Kolb F. Robotic Prophylactic Nipple-Sparing Mastectomy with Immediate Prosthetic Breast Reconstruction: A Prospective Study. Ann Surg Oncol. 2018 Sep;25(9):2579-2586. doi: 10.1245/s10434-018-6555-x. Epub 2018 Jun 29. PMID 29959612
- [Result] Rathat G, Blay L, Bakenga J, Roggen N, Peralta G, Baekelandt J. Scarless preventive surgery. Int J Gynaecol Obstet. 2023 Nov;163(2):701-702. doi: 10.1002/ijgo.15039. Epub 2023 Aug 7. No abstract available. PMID 37548070
- [Result] Rathat G, Fontaine V, Chaumette M, Duraes M. [How I do... an endoscopic mastectomy in 10 steps]. Gynecol Obstet Fertil Senol. 2024 Nov;52(11):653-656. doi: 10.1016/j.gofs.2024.05.004. Epub 2024 May 29. No abstract available. French. PMID 38821450
- [Derived] Rathat G, Chaumette M, Fontaine V, Rebel L, Pissarra J, Duflos C, Duraes M. Endoscopic prophylactic nipple-sparing mastectomy: First French survey of 10 patients. J Gynecol Obstet Hum Reprod. 2025 Jan;54(1):102862. doi: 10.1016/j.jogoh.2024.102862. Epub 2024 Oct 10. PMID 39393530
- See also: Institut national du cancer — http://www.e-cancer.fr/Professionnels-de-sante/Recommandations-et-outils-d-aide-a-la-pratique/Oncogenetique-ou-Cancers-avec-predispositions-genetiques